CLINICAL TRIAL: NCT05987540
Title: Simple, Home-use Neurostimulation tReatment for Parkinson's Disease dEmeNtia
Brief Title: SHARPEN - Parkinson's Disease Dementia
Acronym: SHARPEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company closure
Sponsor: Scion NeuroStim (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS-PD-004; 1R43NS132653-01 (NIH)
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease Dementia
Keywords: medical device; Non-Invasive Brain Stimulation; neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Investigational Treatment (Experimental): Time-varying caloric vestibular stimulation
  Interventions: Device: Non-invasive brainstem stimulation

INTERVENTIONS:
Device: Non-invasive brainstem stimulation — Study participants will self-administer ~19-minute treatments twice daily in the home setting over 12 weeks using a non-invasive brainstem modulation device.

SUMMARY:
The purpose of this single arm study is to evaluate the feasibility and safety of treatments with a non-invasive neuromodulation device in adults diagnosed with mild/moderate Parkinson's disease dementia (PDD). A non-invasive device is a device that stays outside of the body and is not implanted and does not penetrate the skin.

Neuromodulation means that the device stimulates activity in the brain.

DETAILED DESCRIPTION:
Up to 12 participants will self-administer treatments twice daily in the home setting over a period of 12 weeks. There are 4 study center visits, including an eligibility visit, as well as multiple phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 50 years of older, diagnosed with Clinically Established or Clinically Probable Parkinson's disease according to the MDS Clinical Diagnostic Criteria
* Participants with a clinical diagnosis of probable Parkinson's disease dementia ( PDD) using criteria defined in Emre et al., 2007 and in accordance with procedures defined in Dubois et al., 2007 (allowing for diagnosis of PD defined in Step 1 to be according to MDS Clinical Diagnostic criteria instead of the Queen Square Brain Bank Criteria)
* Participants must be able and willing to consent to participate in the study and comply with all study requirements. If the participant is unable to consent due to limited capacity, a Legally Authorized Representative (LAR) must consent.
* Participants and investigators must expect that the participant will be able to remain on a stable regimen of concomitant therapies used for the management of PD and not to introduce new medications used to treat PD (motor or non-motor symptoms) during the study.
* The principal investigator, or designee, must have confidence in the participant's ability to reliably use the TNM™ device, and to understand and complete the assessments (provided in English only) within a given on-state.
* Participant must have a study partner (defined as someone who sees the participant for more than three hours a day, 5 times per week) that is willing to consent and participate in the trial.

Exclusion Criteria:

* Participant anticipates being unable to attend all visits and complete all study activities during the trial.
* Women of child-bearing potential who are pregnant or plan to become pregnant during the course of the trial
* Has any significant co-morbidity/condition, planned surgery or participation in another clinical trial which may either prevent safe participation in the study procedures or interfere with the evaluation of safety or efficacy of the study Device as a potential treatment for PDD
* In the Investigator's opinion, has severe dementia, (e.g., Mini Mental State Exam score (at screen visit) <15 and/or requires significant assistance with activities of daily living due to cognitive deficits)
* Has experienced a myocardial infarction, angina, or stroke within the past 12 months, transient ischemic attack (TIA) within the past 6 months or has a documented aspiration event in the medical records
* Are receiving late-stage therapies for PD (e.g., deep brain stimulation or pump infusion therapies) or are being treated with another neurostimulation device
* History of interventional brain surgery or have received magnetic resonance guided high intensity focused ultrasound
* Demonstrate suicidality at screening (scores ≥ 4 on the Columbia- Suicide Severity Rating Scale Baseline "In the past Month" section)
* Have been previously diagnosed with either clinically meaningful central vestibular dysfunction (lifetime) or have experienced clinically meaningful peripheral vestibular dysfunction within the last 12 months
* Have active ear infections, perforated tympanic membrane or labyrinthitis, as identified by a general ear examination
* Use any drugs excluded in the Excluded Medications List
* Use of antipsychotic medication(s) listed in the Approved Concomitant Medications (i.e., pimavanserin and quetiapine) that have not been taken for more than 180 days and does not have medical record documentation of normal QTc interval (i.e., no prolongation of the QTc interval) as measured via electrocardiogram after starting the medication
* Have active ear infections, perforated tympanic membrane or labyrinthitis, as identified by a general ear examination performed by medically qualified Investigators or have chronic tinnitus that has been ongoing for at least 3 months
* Have a cochlear implant, myringotomy tubes or hearing aids that cannot be easily/reliably removed for treatment
* Clinically significant abnormalities in B12, thyroid function, blood count, comprehensive metabolic panel or urinalysis results tested at the study screen. Screening tests are not required in cases where test results within normal range within 6 months of study screen are documented in the medical records.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of Kansas Medical Center-Parkinson's Disease Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Treatment
Started | 9
Completed | 3
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Study Termination | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 75 [62 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Montreal Cognitive Assessment (MoCA) [Median (Full Range); unit: Total points] — The MoCA assesses cognition over 6 domains: Memory, Executive function, Attention, Language, Visuospatial, and Orientation. Points across all 6 domains are summed, and this sum equals the total score (min 0 - max 30). A higher total score indicates better cognitive function; a positive score for difference in points indicates improvement. A total score of 26-30 reflects normal cognition. Mild cognitive impairment is associated with a total score of 18-25. Total scores of 10 - 17 indicate moderate cognitive impairment; a total score less than 10 shows severe cognitive impairment.
  Total points | 18 [9 to 24]
MDS-UPDRS (Sum of Parts I, II, and III) [Median (Full Range); unit: Total points] — The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates motor (Parts I and III) and non-motor (Part II) experiences and complications of Parkinson's disease (PD) by which it characterizes the extent and burden of disease. Questions/evaluations are divided across Part I (13), Part II (13), Part III (33 scores based on 18 items, several with right, left or other body distribution scores) and summed. Each question has five response options linked to accepted clinical terms: 0/normal, 1/slight, 2/mild, 3/moderate, and 4/severe.
  Total points | 76 [46 to 109]

OUTCOME MEASURES:

1. Primary Outcome: MDS-UPDRS (Sum of Parts I, II & III)
Description: Parts I, II, and III of the International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates motor (Parts I and III) and non-motor (Part II) experiences and complications of Parkinson's disease (PD) by which it characterizes the extent and burden of disease. Questions/evaluations are divided across Part I (13 questions, 52 possible points), Part II (13 questions, 52 possible points), Part III (33 questions based on 18 items, several with right, left or other body distribution scores, 132 possible points) and summed. Each question has five response options linked to accepted clinical terms (0/normal, 1/slight, 2/mild, 3/moderate, and 4/severe) for a total possible score of 236.
  The change between baseline and Day 84 is reported. A positive change in scores between baseline to Day 84 indicates symptom/disease worsening. A negative change in score between baseline and Day 84 indicates symptom/disease improvement.
Time Frame: 12 weeks
Population: Participants that completed an end of treatment visit or early termination visit.
Measure: Median (Full Range); unit: # of points difference
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 5
# of points difference | -2 [-7 to 17]
Statistical Analysis 1: Comparison: Investigational Treatment; Test type: Superiority; p = .8125, Wilcoxon matched-pairs signed rank

2. Primary Outcome: Feasibility of Neuromodulation Device Use in PDD Population, Part 1
Description: Retention rate or the percent of participants that complete the secondary endpoint (MoCA) at all study visits in the study protocol during the 12-week treatment period. High retention: >90%, Moderate retention: 60-90 %, Low retention:< 60 %
Time Frame: 12 weeks
Population: Enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 9
Participants | 3

3. Primary Outcome: Feasibility of Neuromodulation Device Use in PDD Population, Part 2
Description: Treatment adherence rate during the 12-week treatment period. High adherence: >84%, Moderate adherence: 55-84 %, Low adherence: < 55 %
Time Frame: 12 weeks
Population: Participants for whom study devices that had been received by the Sponsor prior to study termination allowing for study device data download.
Measure: Median (Full Range); unit: percentage of treatment adherence
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 6
percentage of treatment adherence | 95.4 [10 to 100]

4. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The MoCA assesses cognition over 6 domains: Memory, Executive function, Attention, Language, Visuospatial, and Orientation. Points across all 6 domains are summed, and this sum equals the total score (min 0 - max 30). A higher total score indicates better cognitive function; a positive score for difference in points indicates improvement. A total score of 26-30 reflects normal cognition. Mild cognitive impairment is associated with a total score of 18-25. Total scores of 10 - 17 indicate moderate cognitive impairment; a total score less than 10 shows severe cognitive impairment.
  The change (difference) in the Montreal Cognitive Assessment (MoCA) total score taken at baseline and, again, at the end of treatment visit (Day 84) after 12 weeks of treatment is reported. A positive change in scores indicates improvement; whereas, a negative change in scores between baseline and Day 84 indicates worsening.
Time Frame: 12 weeks.
Population: Participants that completed the MoCA at the End of Treatment visit (day 84) or early termination visit
Measure: Median (Full Range); unit: # of points difference
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 5
# of points difference | 0 [-4 to 4]
Statistical Analysis 1: Comparison: Investigational Treatment; Test type: Superiority; p > 0.9999, Wilconxon matched-pairs signed rank test

ADVERSE EVENTS:
Time Frame: 4 months, starting with consent.
Description: ct.gov definitions were used.
Groups:
- Investigational Treatment: Time-varying caloric vestibular stimulation (tvCVS)
Arm/Group | Investigational Treatment
All-Cause Mortality (participants affected / at risk) | 1/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=9)
COVID-19 (Infections and infestations) | 2 (2)
Pneumonitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=9)
Device Site Discomfort (Ear and labyrinth disorders) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Difficulty with return of objects (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor company was dissolved prior to completion of participant enrollment. This early termination limited the data analysis to the small number of participants that had completed, prevented completion of treatment adherence data collection from all study devices, and impacted final data close-out activities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT05987540/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT05987540/SAP_001.pdf